CLINICAL TRIAL: NCT04097730
Title: Steroids and Cross-linking for Ulcer Treatment
Acronym: SCUT II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas M. Lietman (Other)
Collaborators: Aravind Eye Care System (Other); National Eye Institute (NEI) (NIH); University of Miami (Other); Stanford University (Other)
Responsible Party: Sponsor-Investigator, Thomas M. Lietman, Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-26045; UG1EY028518 (NIH)
Record Dates: First submitted 2019-09-12; First posted 2019-09-20 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Keratitis Bacterial
MeSH Terms: interventions — Corneal Cross-Linking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Standard Therapy (Placebo Comparator): Participants in this arm will receive topical 0.5% moxifloxacin plus topical placebo plus sham corneal cross-linking.
  Interventions: Drug: Moxifloxacin Ophthalmic; Drug: Riboflavin Ophthalmic; Other: Topical Placebo
- Early Steroids (Experimental): Participants in this arm will receive topical 0.5% moxifloxacin plus topical steroids plus sham corneal cross-linking.
  Interventions: Drug: Moxifloxacin Ophthalmic; Drug: Difluprednate Ophthalmic
- Cross-Linking plus Early Steroids (Experimental): Participants in this group will receive topical 0.5% moxifloxacin plus topical steroids plus corneal cross-linking.
  Interventions: Drug: Moxifloxacin Ophthalmic; Drug: Difluprednate Ophthalmic; Drug: Riboflavin Ophthalmic

INTERVENTIONS:
Drug: Moxifloxacin Ophthalmic — Topical moxifloxacin 0.5% is a fluoroquinolone antibiotic that is used to treat bacterial infections. This is standard therapy for bacterial keratitis. Immediately after CXL/sham CXL and repeat culture, all participants will receive topical moxifloxacin drops every 1 hour for 2 days, and then every 2 hours while awake until resolution of the epithelial defect.
Drug: Difluprednate Ophthalmic — Difluprednate 0.05% is a corticosteroid used to reduce inflammation in the eye. Participants will receive one drop of 0.05% difluprednate four times daily beginning 24 hours after the initiation of antibiotics for 1 week, decreased by 1 drop weekly for a total of 4 weeks of steroid therapy.
  Arms: Cross-Linking plus Early Steroids; Early Steroids
Drug: Riboflavin Ophthalmic — All participants will receive a 30 minute loading dose of topical 0.1% riboflavin and 20% dextran T500 drops every 2 minutes. For participants randomized to corneal cross-linking(CXL), this will be followed by exposure to UV-A light at a wavelength of 365 nm with an irradiance of 3 mW/cm2 for 30 minutes for a total dose of 5.4 J/cm2 (UV lamp: PESCHKE Meditrade GmbH, Hueneberg, Switzerland for India; Avedro KXL System, Waltham, MA, USA for USA). During irradiation patients will continue to receive topical riboflavin at 5-minute intervals. For those randomized to sham CXL, this experience is simulated however the light will be shined adjacent to the patient, careful to avoid exposure to the cornea.
  Other Names: Corneal Cross-Linking with Riboflavin Ophthalmic
  Arms: Cross-Linking plus Early Steroids; Standard Therapy
Other: Topical Placebo — Participants randomized to topical placebo will receive topical placebo on the same medication schedule as difluprednate: one drop of 0.05% difluprednate four times daily beginning 24 hours after the initiation of antibiotics for 1 week, decreased by 1 drop weekly for a total of 4 weeks of placebo therapy. Placebo will be the vehicle used in difluprednate.
  Arms: Standard Therapy

SUMMARY:
Steroids and Cross-linking for Ulcer Treatment (SCUT II) is an international, randomized, double-masked, clinical trial. The purpose of this study is to determine differences in 6-month visual acuity between medical antimicrobial treatments alone versus antimicrobial treatment plus collagen cross-linking (CXL), as well as to further evaluate findings from subgroup analyses of SCUT. Patients presenting to the Aravind Eye Care System (India), Kaiser Permanente Northern California (USA), or the University of California, San Francisco (USA) with smear-positive and/or culture-positive typical (i.e. non-Nocardia or Mycobacteria) bacterial corneal ulcers and moderate to severe vision loss, defined as Snellen visual acuity of 20/40 or worse, will be eligible for inclusion. Those who agree to participate will be randomized to one of three treatment groups:

Group 1: Standard therapy, topical 0.5% moxifloxacin plus topical placebo plus sham CXL Group 2: Early steroids, topical 0.5% moxifloxacin plus topical difluprednate 0.05% plus sham CXL Group 3: CXL plus early steroids, topical 0.5% moxifloxacin plus topical difluprednate 0.05% plus CXL

ELIGIBILITY:
Inclusion Criteria:

* Corneal ulcer that is smear positive and/or culture positive (within 24 hours) for typical bacteria (i.e. non-Nocardia or Mycobacteria)
* Moderate to severe vision loss, defined as Snellen visual acuity of 20/40 (6/12) or worse
* Corneal thickness ≥350 µm, as measured on AS-OCT
* Age over 18 years
* Basic understanding of the study as determined by the physician
* Commitment to return for follow up visits

Exclusion Criteria:

* Evidence of concomitant infection on exam, gram stain, or confocal microscopy (i.e. herpes, both bacteria and acanthameoba on gram stain)
* Impending or frank perforation at recruitment
* Involvement of sclera at presentation
* Non-infectious or autoimmune keratitis
* History of corneal transplantation or recent intraocular surgery
* Pinhole visual acuity worse than 20/200 in the unaffected eye
* Participants who are decisionally and/or cognitively impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2024-05-18 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
Best Spectacle-Corrected Visual Acuity | 6 Months
  Best Spectacle-Corrected Visual Acuity

SECONDARY OUTCOMES:
Best Spectacle-Corrected Visual Acuity | 3 Weeks, 3 Months, 12 Months
  Best Spectacle-Corrected Visual Acuity
Number of Ulcers Testing Positive for Bacteria on Repeat Culture | 2 Days
  Microbiological cure on repeat culture: A scraping of the corneal ulcer taken at 48 hours, then swabbed onto a culture plate and assessed for bacteria
Scar Size | 3 Weeks, 3 Months, 6 Months 12 Months
  Geometric Mean
Scar Depth | 3 Weeks, 3 Months, 6 Months, 12 Months
  Geometric Mean
Adverse Events | 12 Months
  Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Tom Lietman, MD, Principal Investigator — University of California, San Francisco; Jennifer Rose-Nussbaumer, MD, Principal Investigator — Stanford University; Nicole Varnado, MPH, Study Director — Stanford University
Locations (3):
- United States (2):
  - Francis I. Proctor Foundaiton, San Francisco, California
  - University of Miami, Miami, Florida
- Aravind Eye Care System, Madurai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prajna NV, Lalitha P, Chandru S, Radhakrishnan N, Christy J, Karthikeyan A, Rajaraman R, Ramesh R, Amescua G, Mandlik K, Abdelrahman S, Varnado N, Kanchugantla M, Arnold B, Lietman TM, Rose-Nussbaumer JR. Steroids and Cross-Linking for Ulcer Treatment: The SCUT II Randomized Clinical Trial. JAMA Ophthalmol. 2025 Jul 24;143(9):723-30. doi: 10.1001/jamaophthalmol.2025.2188. Online ahead of print. PMID 40705354
- [Derived] Keenan JD. Steroids in the Management of Infectious Keratitis. Cornea. 2023 Nov 1;42(11):1333-1339. doi: 10.1097/ICO.0000000000003340. Epub 2023 Jul 4. PMID 38112645
- [Derived] Radhakrishnan N, Prajna VN, Prajna LS, Venugopal A, Narayana S, Rajaraman R, Amescua G, Porco TC, Lietman TM, Rose-Nussbaumer J. Double-masked, sham and placebo-controlled trial of corneal cross-linking and topical difluprednate in the treatment of bacterial keratitis: Steroids and Cross-linking for Ulcer Treatment Trial (SCUT II) study protocol. BMJ Open Ophthalmol. 2021 Nov 29;6(1):e000811. doi: 10.1136/bmjophth-2021-000811. eCollection 2021. PMID 34901464